CLINICAL TRIAL: NCT04806373
Title: Prospective Randomized Double-Blind Controlled Trial of Intrapleural Fibrinolytic Therapy to Enhance Chemical Pleurodesis
Brief Title: Intrapleural Fibrinolytic Therapy to Enhance Chemical Pleurodesis Enhance Chemical Pleurodesis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Memorial Healthcare System (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MHS 2020.144; ML42028 (Other: Genentech)
Record Dates: First submitted 2021-03-16; First posted 2021-03-19 (Actual); Results first posted 2024-12-11 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Pleural Effusion
MeSH Terms: conditions — Pleural Effusion | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Intervention Model Description: single center, prospective, randomized, double-blind, placebo-controlled trial with two arms
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind. Pharmacist will be unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Talc Slurry Pleurodesis (TSP) plus placebo (Placebo Comparator): Patients who sign informed consent may be randomized to receive TSP alone (talc, 5 gm in 50 ml NS) with placebo (50 ml Normal saline (NS)) through the chest pleural catheter.
  Interventions: Drug: Talc Slurry Pleurodesis
- Talc Slurry Pleurodesis (TSP) plus Cathflo Activase (Experimental): Patients who sign informed consent may be randomized to receive TSP (Talc, 5mg in 50ml Normal saline (NS)) with cathflo activase (4 mg in 50 ml NS) through the chest pleural catheter
  Interventions: Drug: Cathflo Activase; Drug: Talc Slurry Pleurodesis

INTERVENTIONS:
Drug: Cathflo Activase — Cathflo Activase 4mg in 50ml normal saline given through chest pleural catheter
  Arms: Talc Slurry Pleurodesis (TSP) plus Cathflo Activase
Drug: Talc Slurry Pleurodesis — Talc, 5 gm in 50 ml Normal Saline given through chest pleural catheter
  Other Names: TSP

SUMMARY:
Prospective Randomized Double-Blind Controlled Trial of Intrapleural Fibrinolytic Therapy to Enhance Chemical Pleurodesis versus Standard of care Talc therapy in patients with recurrent pleural effusion.

DETAILED DESCRIPTION:
This protocol describes a prospective, randomized, double-blind controlled trial comparing TSP alone to the combination of TSP with cathflo activase for achieving optimal results with pleurodesis for recurrent pleural effusion. Patients who sign informed consent will be randomly assigned to receive either TSP alone (talc, 5 gm in 50 ml NS) with placebo (50 ml NS) or TSP with cathflo activase (4 mg in 50 ml NS) through the chest pleural catheter. Follow-up lasts for three months. The primary outcome is achievement of a "Radiographically Satisfactory Pleurodesis" (RSP) by day three post-procedure, defined as chest tube drainage of less than 100cc over 24 hours and a chest x-ray showing similar or less pleural space opacification than on the day TSP was performed (baseline, day 0). Secondary outcomes include the proportion of patients who achieve RSP, time needed to achieve RSP, duration of chest tube drainage, length of hospital stay after initiation of TSP, proportion of patients requiring repeat TSP, change in serum hemoglobin during therapy, objective assessments of pain and dyspnea, and potential complications. This study will recruit 136 patients, with an interim analyses for efficacy after 50 patients, and aims to help develop the future standard for management of patients requiring pleurodesis for their symptomatic pleural effusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Symptomatic pleural effusion requiring intervention
3. Expected survival > 3 months
4. Written informed consent to trial participation

Exclusion Criteria:

1. Females who are pregnant or lactating
2. Inability to obtain consent from the patient or patient's designated representative.
3. Inability of the patient to comply with the protocol.
4. Previously documented adverse reaction to talc or cathflo activase.
5. Oral or intravenous steroid therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Block, MD, Principal Investigator — Chief, Thoracic Surgery
Locations (1):
- Memorial Healthcare System, Hollywood, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Single center study

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Talc Slurry Pleurodesis (TSP) Plus Placebo | Talc Slurry Pleurodesis (TSP) Plus Cathflo Activase
Started | 12 | 15
Completed | 11 | 14
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Talc Slurry Pleurodesis (TSP) Plus Placebo: Patients who sign informed consent may be randomized to receive talc slurry pleurodesis (TSP) alone (talc, 5 gm in 50 ml NS) with placebo (50 ml Normal saline (NS)) through the chest pleural catheter.
  Talc Slurry Pleurodesis: Talc, 5 gm in 50 ml Normal Saline given through chest pleural catheter
- Talc Slurry Pleurodesis (TSP) Plus Cathflo Activase: Patients who sign informed consent may be randomized to receive talc slurry pleurodesis (TSP) (Talc, 5mg in 50ml Normal saline (NS)) with cathflo activase (4 mg in 50 ml NS) through the chest pleural catheter
  Cathflo Activase: Cathflo Activase 4mg in 50ml normal saline given through chest pleural catheter
  Talc Slurry Pleurodesis: Talc, 5 gm in 50 ml Normal Saline given through chest pleural catheter
- Total: Total of all reporting groups
Arm/Group | Talc Slurry Pleurodesis (TSP) Plus Placebo | Talc Slurry Pleurodesis (TSP) Plus Cathflo Activase | Total
Number analyzed (Participants) | 12 | 15 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (14.5) | 64.6 (15.8) | 65.7 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 12 | 16
  Male | 8 | 3 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 8 | 10 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 11 | 11 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 15 | 27
BMI [Mean (Standard Deviation); unit: kg/m^2] | 23.5 (3.1) | 24.8 (4.5) | 24.2 (3.9)
Effusion etiology [Count of Participants; unit: Participants]
  Lung cancer | 4 | 4 | 8
  Other malignant | 6 | 9 | 15
  Liver disease | 1 | 0 | 1
  Unknown | 1 | 2 | 3
Effusion laterality [Count of Participants; unit: Participants]
  Left | 4 | 3 | 7
  Right | 5 | 10 | 15
  Bilateral | 3 | 2 | 5
Prior pleural intervention [Count of Participants; unit: Participants] | 11 | 14 | 25
Trapped lung [Count of Participants; unit: Participants] | 4 | 8 | 12
Effusion size [Count of Participants; unit: Participants]
  Small (<500 ml) | 8 | 5 | 13
  Moderate (500 - 1000 ml) | 2 | 6 | 8
  Large (>1000 ml) | 2 | 4 | 6
Dyspnea score [Mean (Standard Deviation); unit: units on a scale from 0 to 10, 10 worst] | 0.9 (1.2) | 0.5 (1.5) | 0.7 (1.3)
Chest pain Visual Analog Scale (VAS) [Mean (Standard Deviation); unit: Scale from 0 to 100; with 100 worst pain] | 23.3 (32.4) | 11.9 (28.2) | 17.6 (30.2)

OUTCOME MEASURES:

1. Primary Outcome: Chest X-ray Results on Day 3 After Pleurodesis
Description: Evaluate whether the chest x-ray is better (+1), the same (0), or worse (-1) than it was on the day of pleurodesis
Time Frame: 3-5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Talc Slurry Pleurodesis (TSP) Plus Placebo | Talc Slurry Pleurodesis (TSP) Plus Cathflo Activase
Number analyzed (Participants) | 12 | 15
Participants
  Worse | 5 | 6
  Same | 5 | 8
  Better | 2 | 1
Statistical Analysis 1: Comparison: Talc Slurry Pleurodesis (TSP) Plus Placebo vs Talc Slurry Pleurodesis (TSP) Plus Cathflo Activase; Test type: Other; p = 0.863, Fisher Exact

2. Secondary Outcome: Pleural Drainage Volume (mL) After Pleurodesis
Description: Total volume of drainage on days 1-3 after pleurodesis
Time Frame: 3 days
Measure: Median (Inter-Quartile Range); unit: ml
Arm/Group | Talc Slurry Pleurodesis (TSP) Plus Placebo | Talc Slurry Pleurodesis (TSP) Plus Cathflo Activase
Number analyzed (Participants) | 12 | 15
ml
  Day 1 | 125 [75 to 350] | 427.5 [337.5 to 685]
  Day 2 | 39 [15 to 240] | 150 [55 to 225]
  Day 3 | 45 [0 to 135] | 100 [50 to 200]
Statistical Analysis 1: Comparison: Talc Slurry Pleurodesis (TSP) Plus Placebo vs Talc Slurry Pleurodesis (TSP) Plus Cathflo Activase; Difference in pleural drainage volume day 1 post-TSP; Test type: Other; p = 0.005, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Dyspnea on Day 3 After Pleurodesis
Description: Borg dyspnea scale complete by patient on day 3 after pleurodesis, on a scale of 0 to 10, with 10 being worst.
Time Frame: 3 days
Measure: Median (Inter-Quartile Range); unit: score on a scale from 0 to 10
Arm/Group | Talc Slurry Pleurodesis (TSP) Plus Placebo | Talc Slurry Pleurodesis (TSP) Plus Cathflo Activase
Number analyzed (Participants) | 12 | 15
score on a scale from 0 to 10 | 1 [0 to 3] | 1 [0 to 1.5]
Statistical Analysis 1: Comparison: Talc Slurry Pleurodesis (TSP) Plus Placebo vs Talc Slurry Pleurodesis (TSP) Plus Cathflo Activase; Borg dyspnea scale day 3 post-TSP; Test type: Other; p = 0.891, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Pain Score
Description: Visual analog scale for self-reported level of pain at three days after pleurodesis, from 0 to 100 with 100 being worst pain.
Time Frame: 3 days
Measure: Median (Inter-Quartile Range); unit: score on a scale from 0 to 100
Arm/Group | Talc Slurry Pleurodesis (TSP) Plus Placebo | Talc Slurry Pleurodesis (TSP) Plus Cathflo Activase
Number analyzed (Participants) | 12 | 15
score on a scale from 0 to 100 | 10 [0 to 29.5] | 10 [0 to 30]
Statistical Analysis 1: Comparison: Talc Slurry Pleurodesis (TSP) Plus Placebo vs Talc Slurry Pleurodesis (TSP) Plus Cathflo Activase; Pain score at day 3 post-TSP; Test type: Other; p = 0.899, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Chest Tube Size
Description: Size of the chest tube used for pleural fluid drainage and talc slurry pleurodesis
Time Frame: day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Talc Slurry Pleurodesis (TSP) Plus Placebo | Talc Slurry Pleurodesis (TSP) Plus Cathflo Activase
Number analyzed (Participants) | 12 | 15
Participants
  10 Fr | 4 | 4
  12 Fr | 4 | 4
  14 Fr | 2 | 2
  Unknown | 2 | 5
Statistical Analysis 1: Comparison: Talc Slurry Pleurodesis (TSP) Plus Placebo vs Talc Slurry Pleurodesis (TSP) Plus Cathflo Activase; Test type: Other; p = 0.809, Fisher Exact

6. Secondary Outcome: Time to Chest Tube Removal
Description: Number of days from pleurodesis to removal of the last chest tube
Time Frame: Days from pleurodesis to chest tube removal
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Talc Slurry Pleurodesis (TSP) Plus Placebo | Talc Slurry Pleurodesis (TSP) Plus Cathflo Activase
Number analyzed (Participants) | 12 | 15
days | 7 [5 to 14] | 9 [5 to 12]
Statistical Analysis 1: Comparison: Talc Slurry Pleurodesis (TSP) Plus Placebo vs Talc Slurry Pleurodesis (TSP) Plus Cathflo Activase; Test type: Other; p = 0.946, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Length of Stay
Description: Total duration of hospital stay from admission to discharge, including time before pleurodesis
Time Frame: days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Talc Slurry Pleurodesis (TSP) Plus Placebo | Talc Slurry Pleurodesis (TSP) Plus Cathflo Activase
Number analyzed (Participants) | 12 | 15
days | 10 [6 to 26] | 11 [7 to 15]
Statistical Analysis 1: Comparison: Talc Slurry Pleurodesis (TSP) Plus Placebo vs Talc Slurry Pleurodesis (TSP) Plus Cathflo Activase; Test type: Other; p = 0.808, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Radiographically Satisfactory Pleurodesis
Description: Number (proportion) of patients who achieved daily chest tube drainage of less than 100 cc/24 hours, with the chest x-ray showing no evidence of accumulation of pleural fluid since pleurodesis.
Time Frame: days
Measure: Count of Participants; unit: Participants
Arm/Group | Talc Slurry Pleurodesis (TSP) Plus Placebo | Talc Slurry Pleurodesis (TSP) Plus Cathflo Activase
Number analyzed (Participants) | 12 | 15
Participants | 8 | 12
Statistical Analysis 1: Comparison: Talc Slurry Pleurodesis (TSP) Plus Placebo vs Talc Slurry Pleurodesis (TSP) Plus Cathflo Activase; Test type: Other; p = 0.662, Fisher Exact

9. Secondary Outcome: Time to Achieve Radiographically Satisfactory Pleurodesis
Description: Days from pleurodesis to the point at which pleurodesis is deemed successful and complete
Time Frame: days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Talc Slurry Pleurodesis (TSP) Plus Placebo | Talc Slurry Pleurodesis (TSP) Plus Cathflo Activase
Number analyzed (Participants) | 12 | 15
days | 5.75 (6.27) | 4.83 (3.43)
Statistical Analysis 1: Comparison: Talc Slurry Pleurodesis (TSP) Plus Placebo vs Talc Slurry Pleurodesis (TSP) Plus Cathflo Activase; Test type: Other; p = 0.714, t-test, 2 sided

10. Secondary Outcome: 30 Day Mortality
Description: Number of patients who died within 30 days of pleurodesis
Time Frame: 30 days from pleurodesis
Measure: Number; unit: participants
Arm/Group | Talc Slurry Pleurodesis (TSP) Plus Placebo | Talc Slurry Pleurodesis (TSP) Plus Cathflo Activase
Number analyzed (Participants) | 12 | 15
participants | 4 | 5
Statistical Analysis 1: Comparison: Talc Slurry Pleurodesis (TSP) Plus Placebo vs Talc Slurry Pleurodesis (TSP) Plus Cathflo Activase; Test type: Other; p = 1.0, Fisher Exact

ADVERSE EVENTS:
Time Frame: 60 days
Arm/Group | Talc Slurry Pleurodesis (TSP) Plus Placebo | Talc Slurry Pleurodesis (TSP) Plus Cathflo Activase
All-Cause Mortality (participants affected / at risk) | 4/11 | 5/14
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/14
Other Adverse Events (participants affected / at risk) | 0/11 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/73/NCT04806373/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-09): https://cdn.clinicaltrials.gov/large-docs/73/NCT04806373/ICF_001.pdf